CLINICAL TRIAL: NCT07340892
Title: Prospective Study of NMR-based Serum Metabolic Profiles for the Diagnosis of Checkpoint Inhibitor-related Pneumonitis
Brief Title: Diagnostic Biomarkers for Checkpoint Inhibitor-related Pneumonitis
Status: Recruiting | Type: Observational
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Other Study IDs: CROC202601
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Checkpoint Inhibitor-related Pneumonitis
Keywords: Checkpoint inhibitor-related pneumonitis; ¹H-nuclear magnetic resonance; Metabolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Checkpoint inhibitor-related pneumonitis
- Control group: Lung cancer patients who received immunotherapy but did not develop CIP

SUMMARY:
Checkpoint inhibitor-related pneumonitis (CIP) is a common fatal immune-related adverse events of PD-1/PD-L1 inhibitors. Early diagnosis of CIP is crucial for timely intervention and improved prognosis; however, the absence of precise and effective diagnostic techniques often leads to underdiagnosis and misdiagnosis. The investigators conducted a prospective clinical study to evaluate the effectiveness of ¹H-nuclear magnetic resonance (NMR)-based lipoprotein and metabolite analysis in diagnosing checkpoint inhibitor-related pneumonitis (CIP), aiming to improve its early diagnosis rate.

DETAILED DESCRIPTION:
Checkpoint inhibitor-related pneumonitis (CIP) is a common and potentially fatal immune-related adverse event associated with PD-1/PD-L1 inhibitor therapy. The early and accurate diagnosis of CIP is crucial for timely intervention and improving patient prognosis. However, in clinical practice, the overlapping clinical presentations and imaging features of CIP with infectious pneumonia, tumor progression, or other pulmonary diseases pose a significant diagnostic challenge. The current lack of precise and specific diagnostic techniques often leads to underdiagnosis or misdiagnosis. This diagnostic dilemma can delay the optimal treatment window and may result in the unnecessary interruption or discontinuation of effective immunotherapy, ultimately compromising overall anti-tumor efficacy.

Metabolomics, the comprehensive analysis of small-molecule metabolites, provides a dynamic readout of an organism's physiological state and has shown great promise in biomarker discovery for various diseases. Serum, in particular, offers an easily accessible biofluid that reflects systemic metabolic alterations. ¹H-Nuclear Magnetic Resonance (¹H-NMR) spectroscopy is a robust, reproducible, and quantitative platform ideal for profiling key serum components, including lipoproteins and a wide range of low-molecular-weight metabolites, in a high-throughput manner. The investigators hypothesize that the development of CIP induces a distinct, detectable alteration in the host's systemic metabolic profile, which can be captured by NMR analysis and serve as a diagnostic signature.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathological diagnosis of lung cancer;
2. The subject has received at least one course of immune checkpoint inhibitor treatment;
3. Capable of understanding and voluntarily signing an informed consent form.

   For the CIP group, the following additional criteria must be met:
4. Highly suspected of having checkpoint inhibitor pneumonitis based on radiological abnormalities and/or pulmonary symptoms (including fever, cough, and dyspnea).

   For the Control group, the following additional criteria must be met:
5. Has had no clinical symptoms or radiographic evidence suggestive of pneumonitis at enrollment or prior to enrollment.

Exclusion Criteria:

1. Pulmonary lesions were definitively diagnosed as tumor progression, bacterial pneumonia, or pulmonary edema;
2. Incomplete or missing follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, dual-cohort, biomarker discovery study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | Blood sampling for testing within 1 day after enrollment.
  The Area Under the Receiver Operating Characteristic Curve (AUROC) of a classifier model derived from NMR serum metabolic profiles to distinguish between patients with confirmed checkpoint inhibitor-related pneumonitis and control patients on immunotherapy without pneumonitis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No